CLINICAL TRIAL: NCT02915120
Title: Ultrasound-Guided Pulsed Radiofrequency Of The Genicular Nerves In The Treatment Of Patients With Osteoarthritis Knee Pain: Randomized, Double-Blind, Placebo Controled Trial
Brief Title: Ultrasound-Guided Pulsed Radiofrequency In The Treatment Of Patients With Osteoarthritis Knee (USPRFGENOAK)
Acronym: USPRFGENOAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Javier Mata, Chief of Section of Anesthesiology and Reanimation Department, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RFPGEN-001
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee pain; osteoarthritis; genicular nerve; ultrasonography; pulsed radiofrequency
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Pulsed Radiofrequency (Active Comparator): Before needle insertion, the patient's inferomedial (IM), superomedial (SM), and superolateral (SL) GN branches will be identified under ultrasound guidance. RF needles and probes will be advanced to each of the target nerves under ultrasound guidance. A 50 Hz-frequency sensorial stimulation will be applied with a threshold of < 0.5 mA to identify the nerve position, the current intensity (mA) will be reduced at < 0,2 mA. During the sensorial stimulation, the patients will be asked if they feel tingling, pain, or discomfort inside the knee. The RF probe will be maintained in place until one of those feelings is elicited. In order to avoid inactivating motor nerves, the nerve will be tested for the absence of fasciculation in the the lower extremity on stimulation of 0,5 mA at 2 Hz.
  Interventions: Procedure: Real Pulsed Radiofrequency
- Sham Pulsed Radiofrequency (Sham Comparator): Control patients will undergo the same procedure. The sensorial and motor stimulations will be applied too. The RF electrode will be then inserted through the cannula, and RF lesions will be simulated without applying pulsed RF treatment to the IM, SM and SL, GN branches for 8 minutes each GN branch and the temperature of the electrode tip was not raised.
  Interventions: Procedure: Sham Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Real Pulsed Radiofrequency — Pulsed Radiofrequency uses radiofrequency current in short (20 ms), high-voltage bursts; the "silent" phase (480 ms) allows time for heat elimination, generally keeping the target tissue below 42° C. The Radiofrequency (RF) electrode will be inserted through the canula, and RF lesions will be generated by applying pulsed RF treatment to the inferomedial (IM), superomedial (SM), and superolateral (SL) GN branches for 8 minutes at 42°C.
  Arms: Real Pulsed Radiofrequency
Procedure: Sham Pulsed Radiofrequency — Control patients will undergo the same procedure. The sensorial and motor stimulations will be applied too. The RF electrode will be then inserted through the cannula, and RF lesions will be simulated without applying pulsed RF treatment to the IM, SM and SL, GN branches for 8 minutes each GN branch and the temperature of the electrode tip was not raised.
  Arms: Sham Pulsed Radiofrequency

SUMMARY:
The purpose of this study is to determine if patients with chronic painful knee osteoarthritis experience meaningful and long-term improvement in pain, function, and analgesic use after ultrasound-guided pulsed radiofrequency of the genicular nerves following a double diagnostic genicular nerve blocks.

DETAILED DESCRIPTION:
Osteoarthritis of the knee (kOA) is one of the main causes of disability. Population-based studies revealed that symptomatic kOA is present in 20-30% of the elderly population aged >65 years, and its prevalence is increasing due in part to the aging of the population. The goals of management of patients with kOA are to control pain and to minimize disability. Evidence-based guidelines from National Institute of Health and Clinical Excellence (NICE) and Osteoarthritis Research International (OARSI) suggest that the treatment should be multidisciplinary. Optimal management requires a combination of non-pharmacological (changes in lifestyle, pacing of activities, weight reduction, regular aerobic, acupuncture, muscle strengthening and range of motion exercises) and pharmacological modalities (paracetamol) when additional treatment is required. Total knee arthroplasty (TKA) should be considered for patients with significant symptoms, and/or functional limitations associated with a reduced health-related quality of life, despite conservative therapy. However, there are some fragile patients who are at high risk during surgery and other patients who are not willing to undergo surgery. Because the number of patients will increase as the population ages, alternative approaches to alleviate their joint pain other than conventional treatments are necessary. Ultrasound-guided pulsed radiofrequency of the genicular has recently become a promising treatment option in the management of osteoarthritis related knee pain.

This study is a randomized, double-blind, placebo-controlled trial, parallel design. 142 out-patients with kOA will be recruited from Mallorca, Spain. Participants will be randomly allocated into two groups: Ultrasound-Guided Sham Genicular Nerve Pulsed Radiofrequency without active treatment (Sham GENPRF) and Ultrasound-Guided Real Genicular Nerve Pulsed Radiofrequency (Real GENPRF). All patients will be examined before and 1, 3, 6 and 12 months after the treatment (sham or active).

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain with pain intensity of at least 4 out 10 on the VAS on most or all days for more than 3 months
* Patients of either sex with primary osteoarthritis of one or both knees fulfilling diagnostic criteria for osteoarthritis knee laid down by American College of Rheumatology.
* Patients also had to have a Kellgren-Lawrence (radiologic criterion) score of at least 2
* Pain resistant to conventional therapy including NSAIDs, opioids, muscle relaxants, oral steroids, physical therapy, and intra-articular injection therapy.

Exclusion Criteria:

* The patients with secondary osteoarthritis of knees
* Associated systemic arthropathies, e.g. rheumatoid arthritis and gout
* Previous radiofrequency ablation treatment for similar symptoms.
* Intra-articular knee corticosteroid or hyaluronic acid injection in the past 3 months.
* Active systemic or local infections at the site of proposed needle and electrode placement.
* Coagulopathy or other bleeding disorder
* Cognitive deficit.
* Unstable medical or psychiatric illness.
* Previous knee joint replacement surgery
* Patients missing two or more appointments consecutively were excluded from the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in visual analogue scale (VAS) | baseline and the completion of treatment at 12 weeks
  The VAS is a continuous scale made up of a 100-mm, unmarked, horizontal line, upon which the subject makes a hash mark depending on the amount of pain felt; a mark on the far left of the line indicates "no pain" (score of 0), and a mark to the far right qualifies as "pain as bad as it could be" or "unbearable pain" (score of 100).

SECONDARY OUTCOMES:
Change from Baseline in Goldberg Depression and Anxiety scales | at 1 month
  This consists of two subscales (of nine questions for each scale): an anxiety scale (1-9) and a depression scale (10-18). The first questions for each scale (1-4 and 10-13) are preconditioned questions to determine whether the patient should attempt to answer the rest of the questions of the two subscales. Effectively, at least two questions must be answered affirmatively in the first scale (1-4) for the patient to continue; in the second scale, one answer is sufficient for questions 10-13 for the patient to continue with the rest of the questions. This study will use the Spanish version validated by Montón et al.
Change from Baseline in Goldberg Depression and Anxiety scales | at 3 months
  This consists of two subscales (of nine questions for each scale): an anxiety scale (1-9) and a depression scale (10-18). The first questions for each scale (1-4 and 10-13) are preconditioned questions to determine whether the patient should attempt to answer the rest of the questions of the two subscales. Effectively, at least two questions must be answered affirmatively in the first scale (1-4) for the patient to continue; in the second scale, one answer is sufficient for questions 10-13 for the patient to continue with the rest of the questions. This study will use the Spanish version validated by Montón et al.
Change from Baseline in Goldberg Depression and Anxiety scales | at 6 months
  This consists of two subscales (of nine questions for each scale): an anxiety scale (1-9) and a depression scale (10-18). The first questions for each scale (1-4 and 10-13) are preconditioned questions to determine whether the patient should attempt to answer the rest of the questions of the two subscales. Effectively, at least two questions must be answered affirmatively in the first scale (1-4) for the patient to continue; in the second scale, one answer is sufficient for questions 10-13 for the patient to continue with the rest of the questions. This study will use the Spanish version validated by Montón et al.
Change from Baseline in Goldberg Depression and Anxiety scales | up to 1 year
  This consists of two subscales (of nine questions for each scale): an anxiety scale (1-9) and a depression scale (10-18). The first questions for each scale (1-4 and 10-13) are preconditioned questions to determine whether the patient should attempt to answer the rest of the questions of the two subscales. Effectively, at least two questions must be answered affirmatively in the first scale (1-4) for the patient to continue; in the second scale, one answer is sufficient for questions 10-13 for the patient to continue with the rest of the questions. This study will use the Spanish version validated by Montón et al.
Change from baseline in WOMAC index | at 1 month
  The WOMAC scale is used to evaluate the condition of patients with OA of the knee and the hip and includes pain, stiffness, and physical functioning of the joints. This scale measures five items for pain (with a score range of 0-20), two for stiffness (score range of 0-8), and 17 for functional limitation (score range of 0-68). The physical functioning questions cover everyday activities. These scales will be used separately and will not be summed. Patients will respond orally to the five levels with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are left unanswered, the scale will be declared invalid. If the patient does not respond to one question, a mean will be taken from the results of the other questions. The range will be 0-98.
Change from baseline in WOMAC index | at 3 months
  The WOMAC scale is used to evaluate the condition of patients with OA of the knee and the hip and includes pain, stiffness, and physical functioning of the joints. This scale measures five items for pain (with a score range of 0-20), two for stiffness (score range of 0-8), and 17 for functional limitation (score range of 0-68). The physical functioning questions cover everyday activities. These scales will be used separately and will not be summed. Patients will respond orally to the five levels with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are left unanswered, the scale will be declared invalid. If the patient does not respond to one question, a mean will be taken from the results of the other questions. The range will be 0-98.
Change from baseline in WOMAC index | at 6 months
  The WOMAC scale is used to evaluate the condition of patients with OA of the knee and the hip and includes pain, stiffness, and physical functioning of the joints. This scale measures five items for pain (with a score range of 0-20), two for stiffness (score range of 0-8), and 17 for functional limitation (score range of 0-68). The physical functioning questions cover everyday activities. These scales will be used separately and will not be summed. Patients will respond orally to the five levels with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are left unanswered, the scale will be declared invalid. If the patient does not respond to one question, a mean will be taken from the results of the other questions. The range will be 0-98.
Change from baseline in WOMAC index | up to 1 year
  The WOMAC scale is used to evaluate the condition of patients with OA of the knee and the hip and includes pain, stiffness, and physical functioning of the joints. This scale measures five items for pain (with a score range of 0-20), two for stiffness (score range of 0-8), and 17 for functional limitation (score range of 0-68). The physical functioning questions cover everyday activities. These scales will be used separately and will not be summed. Patients will respond orally to the five levels with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are left unanswered, the scale will be declared invalid. If the patient does not respond to one question, a mean will be taken from the results of the other questions. The range will be 0-98.
EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire Changes in baseline use of medication | at 1 month
  This questionnaire will have four questions developed according the EUROHIS (European Health Interview Survey) recommendations in order to harmonize the information regarding medicine use [31]. Subjects will be asked (1) about the prescription medicine their general practitioner may have prescribed for them ("Have you taken any pain medicine prescribed by your general practitioner?") as well as any medication not prescribed by their general practitioner ("Have you taken any pain medicine not prescribed by your general practitioner") and (2) whether or not their prescribed and non-prescribed pain medication use has increased or decreased.
EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire Changes in baseline use of medication | at 3 months
  This questionnaire will have four questions developed according the EUROHIS (European Health Interview Survey) recommendations in order to harmonize the information regarding medicine use [31]. Subjects will be asked (1) about the prescription medicine their general practitioner may have prescribed for them ("Have you taken any pain medicine prescribed by your general practitioner?") as well as any medication not prescribed by their general practitioner ("Have you taken any pain medicine not prescribed by your general practitioner") and (2) whether or not their prescribed and non-prescribed pain medication use has increased or decreased.
EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire Changes in baseline use of medication | at 6 months
  This questionnaire will have four questions developed according the EUROHIS (European Health Interview Survey) recommendations in order to harmonize the information regarding medicine use [31]. Subjects will be asked (1) about the prescription medicine their general practitioner may have prescribed for them ("Have you taken any pain medicine prescribed by your general practitioner?") as well as any medication not prescribed by their general practitioner ("Have you taken any pain medicine not prescribed by your general practitioner") and (2) whether or not their prescribed and non-prescribed pain medication use has increased or decreased.
EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire Changes in baseline use of medication | up to 1 year
  This questionnaire will have four questions developed according the EUROHIS (European Health Interview Survey) recommendations in order to harmonize the information regarding medicine use [31]. Subjects will be asked (1) about the prescription medicine their general practitioner may have prescribed for them ("Have you taken any pain medicine prescribed by your general practitioner?") as well as any medication not prescribed by their general practitioner ("Have you taken any pain medicine not prescribed by your general practitioner") and (2) whether or not their prescribed and non-prescribed pain medication use has increased or decreased.
Change from baseline in a visual analogue scale (VAS) | at 1 month
  The VAS is a continuous scale made up of a 100-mm, unmarked, horizontal line, upon which the subject makes a hash mark depending on the amount of pain felt; a mark on the far left of the line indicates "no pain" (score of 0), and a mark to the far right qualifies as "pain as bad as it could be" or "unbearable pain" (score of 100).
Change from baseline in a visual analogue scale (VAS) | at 6 months
  The VAS is a continuous scale made up of a 100-mm, unmarked, horizontal line, upon which the subject makes a hash mark depending on the amount of pain felt; a mark on the far left of the line indicates "no pain" (score of 0), and a mark to the far right qualifies as "pain as bad as it could be" or "unbearable pain" (score of 100).
Change from baseline in a visual analogue scale (VAS) | up to 1 year
  The VAS is a continuous scale made up of a 100-mm, unmarked, horizontal line, upon which the subject makes a hash mark depending on the amount of pain felt; a mark on the far left of the line indicates "no pain" (score of 0), and a mark to the far right qualifies as "pain as bad as it could be" or "unbearable pain" (score of 100).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mata, MD, Principal Investigator — Son Llatzer University Hospital
Locations (1):
- Son Llatzer University Hospital, Palma, Balear Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
No later than 3 years after the study will have ended a completely deidentified data set will deliver to an appropriate data archive for sharing purposes
Supporting Information: Study Protocol, ICF
Time Frame: Study Protocol, Statistical Analisis Plan and Informed Consent Form will be published in BMJ Open by the end of this year.
  No later than 3 years after the study will have ended a completely deidentified data set will deliver to an appropriate data archive for sharing purposes
Access Criteria: Anyone can get access to the data with no registration or condition (BMJ Open).

REFERENCES:
- [Background] Rubinstein SM, van Tulder M. A best-evidence review of diagnostic procedures for neck and low-back pain. Best Pract Res Clin Rheumatol. 2008 Jun;22(3):471-82. doi: 10.1016/j.berh.2007.12.003. PMID 18519100
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. PM R. 2014 Apr;6(4):373-6. doi: 10.1016/j.pmrj.2013.10.003. Epub 2013 Dec 27. PMID 24373908
- [Background] Masala S, Fiori R, Raguso M, Morini M, Calabria E, Simonetti G. Pulse-dose radiofrequency for knee osteoartrithis. Cardiovasc Intervent Radiol. 2014 Apr;37(2):482-7. doi: 10.1007/s00270-013-0694-z. Epub 2013 Aug 14. PMID 23942592
- [Background] Kesikburun S, Yasar E, Uran A, Adiguzel E, Yilmaz B. Ultrasound-Guided Genicular Nerve Pulsed Radiofrequency Treatment For Painful Knee Osteoarthritis: A Preliminary Report. Pain Physician. 2016 Jul;19(5):E751-9. PMID 27389118
- [Background] Vas L, Pai R, Khandagale N, Pattnaik M. Pulsed radiofrequency of the composite nerve supply to the knee joint as a new technique for relieving osteoarthritic pain: a preliminary report. Pain Physician. 2014 Nov-Dec;17(6):493-506. PMID 25415774
- [Background] Ikeuchi M, Ushida T, Izumi M, Tani T. Percutaneous radiofrequency treatment for refractory anteromedial pain of osteoarthritic knees. Pain Med. 2011 Apr;12(4):546-51. doi: 10.1111/j.1526-4637.2011.01086.x. Epub 2011 Apr 4. PMID 21463469
- [Background] Cosman ER Jr, Dolensky JR, Hoffman RA. Factors that affect radiofrequency heat lesion size. Pain Med. 2014 Dec;15(12):2020-36. doi: 10.1111/pme.12566. Epub 2014 Oct 14. PMID 25312825
- [Background] Yasar E, Kesikburun S, Kilic C, Guzelkucuk U, Yazar F, Tan AK. Accuracy of Ultrasound-Guided Genicular Nerve Block: A Cadaveric Study. Pain Physician. 2015 Sep-Oct;18(5):E899-904. PMID 26431143
- [Background] Kvarstein G. A new target for radiofrequency neurotomy? Pain. 2011 Mar;152(3):465-466. doi: 10.1016/j.pain.2010.09.037. Epub 2010 Oct 18. No abstract available. PMID 20961686
- [Background] Lin ML, Lin MH, Fen JJ, Lin WT, Lin CW, Chen PQ. A comparison between pulsed radiofrequency and electro-acupuncture for relieving pain in patients with chronic low back pain. Acupunct Electrother Res. 2010;35(3-4):133-46. doi: 10.3727/036012910803860940. PMID 21319602
- [Background] Bhatia A, Peng P, Cohen SP. Radiofrequency Procedures to Relieve Chronic Knee Pain: An Evidence-Based Narrative Review. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):501-10. doi: 10.1097/AAP.0000000000000414. PMID 27281721
- [Background] Manzano D, Jimenez F, Blasi M. Ultrasound-guided pain interventions in the knee region. Techniques in Regional Anesthesia and Pain Management. 2013;17:131-9.
- [Background] Franco CD, Buvanendran A, Petersohn JD, Menzies RD, Menzies LP. Innervation of the Anterior Capsule of the Human Knee: Implications for Radiofrequency Ablation. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):363-8. doi: 10.1097/AAP.0000000000000269. PMID 26066383
- [Derived] Mata J, Valenti P, Hernandez B, Mir B, Aguilar JL. Study protocol for a randomised controlled trial of ultrasound-guided pulsed radiofrequency of the genicular nerves in the treatment of patients with osteoarthritis knee pain. BMJ Open. 2017 Nov 3;7(11):e016377. doi: 10.1136/bmjopen-2017-016377. PMID 29102985